CLINICAL TRIAL: NCT05100784
Title: The Human Sperm Survival Assay (HSSA) as an Internal Quality Control for the IVF Consumables
Brief Title: The Human Sperm Survival Assay (HSSA) as an Internal Quality Control for the IVF Consumables (REPROTOX 2)
Acronym: REPROTOX 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other); Private hospital Parly II (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A01972-37
Record Dates: First submitted 2021-10-28; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Human Sperm Survival Assay; Embryotoxicity; in Vitro Fertilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sperm with normal spermogramm and more than 10 millions spermatozoids: Normal spermogramm : concentration ≥15 million / ml or total count> 39 million, progressive mobility ≥32% or total mobility ≥40%
  Interventions: Biological: HSSA test

INTERVENTIONS:
Biological: HSSA test — Human Sperm Survival Assay testing performed on different batches of different types of IVF consumables. In practice, 3 consumables from the same batch will be tested with 3 different sperms to ensure the repeatability of the result / test.

SUMMARY:
The main embryotoxicity quality controls are the mouse embryo test (MEA = Mouse Embryo Assay) and the human sperm survival test (HSSA = Human Sperm Survival Assay). The HSSA test measures the survival (or mobility) of human sperm after exposure to the tested consumable for a predetermined period of time and compares it to that of unexposed sperm. It would appear that the HSSA is comparable in terms of sensitivity to the MEA test for the detection of toxicity.

DETAILED DESCRIPTION:
The main objective is to assess the embryotoxicity of the main IVF consumables using the HSSA test before their introduction to the IVF laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Male over 18 years-old
* Normal spermogram (concentration ≥15 million / ml or total count> 39 million, progressive mobility ≥32% or total mobility ≥40%)
* Progressive mobility ≥70% after selection
* Total number of progressive motile spermatozoa recovered after TMS> 10 million
* Patient affiliated or beneficiary of a social security scheme
* Patient having been informed and not opposing to this research.

Exclusion Criteria:

* Male over 65 years-old
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male between 18 and 65 years-old with normal spermogram
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2022-03-04 (Estimated)

PRIMARY OUTCOMES:
Presence of embryotoxicity | 1 day
  Presence of embryotoxicity, defined by a mobility index relative to the control (SMI) <0.85 observed on at least 2 of the three tests carried out on consumables from the same batch (isolated embryotoxicity).

CONTACTS AND LOCATIONS:
Locations (1):
- Private Hospital of Parly II-Le Chesnay, Le Chesnay, France